CLINICAL TRIAL: NCT02534493
Title: Safety and Efficacy of a Novel Carpal Tunnel Tissue Manipulation Device in Treating Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pressure Profile Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPS-CTMD-15-001
Record Dates: First submitted 2015-03-25; First posted 2015-08-27 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carpal Tunnel Medical Device (CTMD) (Experimental): Carpal Tunnel Tissue Manipulation Device (CTMD)
  Interventions: Device: Carpal Tunnel Tissue Manipulation Device (CTMD)

INTERVENTIONS:
Device: Carpal Tunnel Tissue Manipulation Device (CTMD) — This piece of rigid, shaped, biocompatible plastic (polypropylene) rated for skin contact and a strong but safe hypoallergenic biocompatible medical adhesive which bonds the skin over the carpal tunnel to the plastic piece for a duration of 2-14 hours.
  Other Names: Wrist-Aid

SUMMARY:
A single-center, prospective, non-randomized study to evaluate the safety and efficacy of a novel carpal tunnel tissue manipulation device in treating symptoms and decreased physical function in subjects previously diagnosed with mild to severe carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
A single-center, prospective, non-randomized study to evaluate the safety and efficacy of a novel carpal tunnel tissue manipulation device in treating symptoms and decreased physical function in subjects previously diagnosed with mild to severe carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria

1. male or female, ages 21-65 and in good general health;
2. subject diagnosed with mild to severe carpal tunnel syndrome (CTS) (AANEM criteria for CTS)

   * mild CTS: prolonged distal sensory latency with ± decreased sensory amplitude
   * moderate CTS: abnormal median sensory latency with prolongation of the distal motor latency
   * severe CTS: prolonged motor and sensory distal peak latencies either with a low or absent SNAP or CMAP
3. bilateral CTS accepted (either mild, moderate or severe CTS bilaterally), however, more involved wrist (via NCS) used as "study" wrist;
4. Boston Carpal Tunnel Questionnaire (BCTQ) Symptoms Score ≥ 2;
5. women of childbearing potential must be willing to practice effective contraception for the duration of the study (i.e., abstinence, condoms or diaphragm with spermicide, IUD, or birth control pills [BCP]);

   NOTE: Females on birth control pills (BCP) must be stable on the same type and dose of pill for at least three months prior to entering the study and must not change the type of BCP or dosing regimen during the study. Those who have discontinued using BCPs in favor of another form of contraception must have discontinued BCP usage at least 3 months prior to the start of the study.
6. women of child bearing potential must have a negative urine pregnancy test at the Baseline Visit (Visit 1, Day 0) and must not be lactating; and
7. willingness to follow protocol requirements, including signing an informed consent and health information release forms, attending routine follow-up visits and completing questionnaires.

Exclusion Criteria

1. known sensitivity to adhesives or glue;
2. history of diabetes mellitus;
3. history of thyroid disease;
4. history of prior wrist fractures;
5. known to be easily bruised (hematoma);
6. concurrent use of blood thinners;
7. history of connective tissue disease;
8. diagnosed with superimposed peripheral neuropathy;
9. history of cervical radiculopathy;
10. diagnosed with purely ulnar paresthesias;
11. history of ulnar neuropathy;
12. history of brachial plexopathy;
13. diagnosed with pronator teres syndrome;
14. history of polyneuropathy;
15. uncontrolled systemic disease;
16. history of any mass, tumor, severe trauma or deformity of the hand or wrist;
17. previous surgery of the hand or wrist;
18. history of prior carpal tunnel release;
19. current use of any splinting or bracing medical device for CTS;
20. currently taking any medication therapy that could cause a focal or generalized neuropathy (e.g., antiepileptics, statins, chemotherapeutic or antiarrhythmic);
21. history of any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results;
22. concomitant use of systemic medication(s) or therapy that may have a substantial effect on CTS condition, unless such medication(s) or therapy has/have been used for a minimum of 3 months prior to study enrollment, is/are expected to remain constant throughout the course of the study and is/are considered necessary for a subjects' welfare;
23. females who are pregnant, nursing, or planning a pregnancy or who are of childbearing potential and not using a reliable method of contraception;
24. inability to give informed consent; and
25. concurrent participation or prior participation in any investigation drug or device study within the last 30 days prior to the Baseline Visit (Visit 1).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank J. King, M.D., Principal Investigator — Mission Pain and Spine
Locations (1):
- Mission Pain and Spine, Mission Viejo, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only enrolled if a nerve conduction study (NCS) was performed at the enrollment visit or within the past 6 months, electrodiagnostically confirming the presence of mild to severe CTS.
Units Other Than Participants: per affected wrist
Groups:
- Carpal Tunnel Medical Device (CTMD): The Carpal Tunnel Tissue Manipulation Device (CTMD) is a piece of rigid, shaped, biocompatible plastic (polypropylene) rated for skin contact and a strong but safe hypoallergenic biocompatible medical adhesive which bonds the skin over the carpal tunnel to the plastic piece. The CTMD is worn for a duration of 8-10 hours daily over the treatment period.
  If a participant had bilateral CTS, both wrists were treated but only the worst wrist (via NCS and BCTQ SSS score) was analyzed.
Period: Overall Study
Arm/Group | Carpal Tunnel Medical Device (CTMD)
Started | 13; 19 per affected wrist
Completed | 11; 15 per affected wrist
Not Completed | 2; 4 per affected wrist
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Only the affected wrist was treated in participants with unilateral CTS. Both wrists were treated on participants with bilateral CTS but only the worse wrist (higher severity via NCS or higher BCTQ SSS score) was used for analysis.
Arm/Group | Carpal Tunnel Medical Device (CTMD)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The categories for race and ethnicity were combined, such that the Hispanic choice was lumped with Asian, Caucasian, Black, and Other. The single participant that identified as Hispanic was lumped in with Caucasian in the Race section.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 10
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The categories for race and ethnicity were combined, such that the Hispanic choice was lumped with Asian, Caucasian, Black, and Other. The single participant that identified as Hispanic was lumped in with Caucasian in the Race section.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 8
    More than one race | 0
    Unknown or Not Reported | 0
Bilaterality [Count of Participants; unit: Participants] — Participants presented with either unilateral CTS (only one wrist affected) or bilateral CTS (both wrists affected).
  Participants
    Unilateral CTS | 7
    Bilateral CTS | 4
Severity [Count of Participants; unit: Participants] — Severity determined using a shortened nerve conduction study protocol and using AANEM criteria.
  Participants
    Mild | 3
    Moderate | 4
    Severe | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in SSS of the BCTQ at 28 Days vs Baseline
Description: The primary efficacy variable is the decrease in Symptom Severity Scale (SSS) score of the Boston Carpal Tunnel Questionnaire (BCTQ). The SSS is a patient-reported measure of the severity of the patient's symptoms caused by carpal tunnel syndrome, on a scale of 1 (no symptoms) to 5 (worst symptoms).
Time Frame: 28 days
Population: Primary outcome measures were analyzed for unilateral and bilateral subjects combined, but measures were analyzed for unilateral and bilateral subjects separately as well.
Measure: Mean (Standard Deviation); unit: point decrease in SSS
Groups:
- Unilateral+Bilateral: The CTMD was worn for a duration of 8-10 hours daily over the treatment period. Unilateral subjects wore the CTMD on the single affected wrist. Bilateral subjects wore the CTMD on both wrists, but only the worst wrist (via NCS and BCTQ SSS score) was analyzed.
- Unilateral Only: The CTMD was worn for a duration of 8-10 hours daily over the treatment period. Unilateral subjects wore the CTMD on the single affected wrist.
- Bilateral Only: The CTMD was worn for a duration of 8-10 hours daily over the treatment period. Bilateral subjects wore the CTMD on both wrists, but only the worst wrist (via NCS and BCTQ SSS score) was analyzed.
Arm/Group | Unilateral+Bilateral | Unilateral Only | Bilateral Only
Number analyzed (Participants) | 11 | 7 | 4
point decrease in SSS | 0.59 (0.68) | 0.93 (0.52) | .00 (0.50)

2. Secondary Outcome: Change in SSS of the BCTQ 2 Month Post-treatment vs Baseline
Description: The secondary efficacy variable is the decrease in Symptoms Severity Scale (SSS) score of the Boston Carpal Tunnel Questionnaire (BCTQ) obtained 2 months after the 28-day CTMD treatment period compared to the Baseline SSS score.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: point decrease in SSS
Arm/Group | Unilateral+Bilateral | Unilateral Only | Bilateral Only
Number analyzed (Participants) | 11 | 7 | 4
point decrease in SSS | 0.79 (0.74) | 1.20 (0.53) | 0.09 (0.41)

ADVERSE EVENTS:
Time Frame: 3 months (1 month device wear and 2 months post-treatment) per subject
Description: Inclusion of Unanticipated Adverse Device Event (ADE) in addition to SAE, to clarify serious adverse events caused by associated with the device.
  Adverse events self-reported by subjects and recorded in AE logs.
Arm/Group | Carpal Tunnel Medical Device (CTMD)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carpal Tunnel Medical Device (CTMD) (N=11)
Skin Reddening/Irritation (Skin and subcutaneous tissue disorders) | 7 — reddening, itching, and minor irritation of skin due to contact with adhesive and pull from device
Acute Irritation (Product Issues) | 2 — Edge of device pressed into subjects' wrists, causing acute but minor pain

LIMITATIONS AND CAVEATS:
This study was an open-label pilot study with no placebo. Subjects were not allowed other CTS treatments except for occasional painkillers. Daily home activities not controlled. One subject had wrist arthritis. One subject had unconfirmed arthritis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No